CLINICAL TRIAL: NCT03550833
Title: Impact of Life Events and Psychological Stress in Rheumatoid Arthritis Set-up : Case-control Study Within a Multifactorial and Integrative Psychological Model
Acronym: Stress-PR
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/01
Record Dates: First submitted 2018-05-28; First posted 2018-06-08 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Arthritis, Rheumatoid; Stress Disorder
Keywords: Rheumatoid arthritis; Stress
MeSH Terms: conditions — Arthritis, Rheumatoid; Stress Disorders, Traumatic | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rheumatoid Arthritis patients: patients affected by RA according to ACR/EULAR 2010 criteria, with a disease duration less than 2 years
  Interventions: Behavioral: Questionnaire; Biological: blood sample
- control patients: patients with a visceral surgery for less than 2 years (appendectomy, cholecystectomy, bowel obstruction, hernia, eventration…)
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire
Biological: blood sample — 7 ml whole blood for Peripheral blood
  Groups: Rheumatoid Arthritis patients

SUMMARY:
Rheumatoid Arthritis (RA) is an inflammatory rheumatic disease that can lead to structural damage and handicap. The RA physiopathology is multifactorial, including genetic and environmental risk factors. The identification of environmental factors implication is crucial to understand the RA mechanism, and improves the diagnosis and the treatment of the disease.

DETAILED DESCRIPTION:
The physiopathology of RA is multifactorial, implicating genetic and environmental factors. Within the environmental factors, the exact role of psychological stress and life events on the onset of the disease is still under question. In clinical practice, patients usually report the occurrence of a stressing life event before the diagnosis of the disease (mourning, dismissal, divorce…). Nevertheless, literature reviews present some discrepancies and did not lead to a clear identification of the role of psychological stress in RA onset. This is mainly due to the evaluation methods of stress within those previous studies, considering stress as a unique response of the organism without taking into account personal, sociological, biological or environmental history. The aim of the study is to analyze the impact of stress on the RA onset within an integrative model, to evaluate patient assessment of the stress, and to present strategies to fix it.

ELIGIBILITY:
Patients RA :

Inclusion Criteria:

* patients aged over 18 years old
* patients affected by RA according to ACR/EULAR 2010 criteria, with a disease duration less than 2 years.
* Speaking and understanding French language
* Being informed about the study and having given his oral consent

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patient who refuse to participate.

Control :

Inclusion Criteria:

* patients aged over 18 years old
* patients with a visceral surgery for less than 2 years (appendectomy, cholecystectomy, bowel obstruction, hernia, eventration…)
* Speaking and understanding French language
* Being informed about the study and having given his oral consent

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patient who refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by RA according to ACR/EULAR 2010 criteria, with a disease duration less than 2 years
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
Life events calculated over the year preceding the onset of PR symptoms | At inclusion (day 0)
  Social Readjustment Rating Scale (SRRS)

SECONDARY OUTCOMES:
Perceived stress | At inclusion (day 0)
  Perceived Stress Scale (PSS)
Perceived control | At inclusion (day 0)
  Multidimensional Health Locus of Control Scale (MHLCS)
Perceived social support | At inclusion (day 0)
  Social Support Questionnaire (SSQ)
State Anxiety | At inclusion (day 0)
  State-Trait Anxiety Inventory (STAI-Y-A)
Coping | At inclusion (day 0)
  Ways of Coping Checklist Scale (WCC)
Cytokine levels in RA patients sera | 12 months from baseline
Correlation between cytokine levels and RA activity | 12 months from baseline
Correlation between cytokine levels and stress for RA patients | 12 months from baseline
Identification of neuropathic pain for RA patients evalued by douleur-neuropathique 10 items questionnaire | 12 months from baseline
  douleur-neuropathique 10 items questionnaire providing a score between 0 and 10, with a positive threshold value beyond 4/10.
Characterization of neuropathic pain for RA patients evalued by Neuropathic Pain Symptom Inventory questionnaire | 12 months from baseline
  Neuropathic Pain Symptom Inventory questionnaire with 12 items to complete, providing for each item the presence (or the absence) of several pain symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Thierry SCHAEVERBEKE, Prof, Principal Investigator — University Hospital, Bordeaux
Locations (5):
- France (5):
  - CHU de Bordeaux - service de rhumatologie, Bordeaux
  - CH de Dax - service de rhumatologie, Dax
  - Hôpital Suburbain du Bouscat, Le Bouscat
  - CH de Libourne - service de rhumatologie, Libourne
  - CH de Pau - service de rhumatologie, Pau